CLINICAL TRIAL: NCT04780867
Title: The Influence of Psychosocial and Lifestyle Factors on Immune Health and Injury Incidence During Phase One Training in UK Army Recruits
Brief Title: Psychological and Lifestyle Factors on Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Nottingham (Other); University of California, Los Angeles (Other); Loughborough University (Other); Ministry of Defence, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1070/MODREC/20
Record Dates: First submitted 2021-02-15; First posted 2021-03-04 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-04

CONDITIONS: Psychological; Stress; Immune Health; Vaccination; Respiratory Tract Infections; Injury
MeSH Terms: conditions — Respiratory Tract Infections; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: For aim 1, an observational design will be used to examine the influence of psychosocial and lifestyle factors at the start of basic Army training on immune health (e.g. respiratory infection and antibody response to influenza vaccination) and injury during training.
  For aim 2, the recruited cohort will be divided into two groups: (i) Routine vaccination group: to receive first hepatitis B vaccination at initial medical assessment upon entry to basic training and second hepatitis B vaccination 1 month later; (ii) Delayed vaccination group: to receive first hepatitis B vaccination during week 5 of training and second hepatitis B vaccination 1 month later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine vaccination (Control) (No Intervention)
- Delay vaccination (Experimental) (Experimental)
  Interventions: Behavioral: Delayed vaccination

INTERVENTIONS:
Behavioral: Delayed vaccination — First and second hepatitis B vaccinations will be delayed by 1 month in the interventional group to establish whether changes in psychosocial and lifestyle factors during training impact immune health.
  Arms: Delay vaccination (Experimental)

SUMMARY:
Psychosocial and lifestyle factors in Army recruits likely contribute to increased susceptibility to infection and injury during basic Army training. The primary aim of this study is to assess the influence of psychosocial and lifestyle factors at the start of basic Army training on immune health (e.g. respiratory infection and antibody response to influenza vaccination) and injury during training, in an observational design.

A secondary aim is to establish whether changes in psychosocial and lifestyle factors during training impact immune health (e.g. response to hepatitis B vaccination). Using an interventional design, participants will be randomly allocated into two experimental groups: (i) Routine vaccination group: to receive first hepatitis B vaccination at initial medical assessment upon entry to basic training and second hepatitis B vaccination 1 month later; (ii) Delayed vaccination group: to receive first hepatitis B vaccination during week 5 of training and second hepatitis B vaccination 1 month later.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 16-33 years enrolled in phase one British Army training

Exclusion Criteria:

-

Ages: 16 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1188 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Antibody response to influenza vaccination - Aim 1 | 1 month
Physician diagnosed respiratory infection incidence - Aim 1 | 6 months
Physician diagnosed injury incidence - Aim 1 | 6 months
Antibody response to second hepatitis B vaccination - Aim 2 | Routine group: 3 months; Delay group: 4 months

SECONDARY OUTCOMES:
Antibody response to influenza vaccination | 4 months
Antibody response to first hepatitis B vaccination | Routine group: 1 months; Delay group: 2 months
C-reactive protein | Baseline, 1-day post vaccination and 1 month
Gene expression profiling | Baseline and 1 month
Epstein Barr Virus serostatus/antibody titre | Baseline and 1 month
Cytomegalovirus serostatus/antibody titre | Baseline and 1 month
Torque Teno Virus plasma DNA | Baseline and 1 month
Interleukin-6 | Baseline and 1 month
Hair cortisol | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Walsh, PHD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Infantry Training Centre, Catterick, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No